CLINICAL TRIAL: NCT03292549
Title: RObotic PArtial Nephrectomy National Study (RoPaN Study)
Brief Title: RObotic PArtial Nephrectomy National Study
Acronym: ROPAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/30
Record Dates: First submitted 2016-07-12; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2016-07

CONDITIONS: Kidney Cancer
Keywords: Urology; Robotic surgery; Haemostasis; Partial Nephrectomy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Robotic partial surgery
  Interventions: Procedure: Robotic partial surgery

INTERVENTIONS:
Procedure: Robotic partial surgery — Robotic partial surgery

SUMMARY:
The purpose of the study is to set up the larger prospective study on robotic partial nephrectomy, to describe the characteristics of patients operated for kidney cancer by this surgical procedure and also to determine the modalities of hemostasis in this procedure.

DETAILED DESCRIPTION:
The primary objective of the study is to describe the characteristics of patients operated for kidney cancer by a robotic partial nephrectomy in France (recruiting centers, patient profile, tumor characteristics).

Secondary Objective(s):

1. To describe the surgical techniques and operative development.
2. To assess the modalities of haemostasis, during robotic partial nephrectomy.
3. To assess peri-operative morbidity in robotic partial nephrectomy and post-operative complications.
4. To assess the outcome of renal function after a robotic partial nephrectomy. This study is a national, multicenter, prospective, cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old at the time of screening
* Subject has been diagnosed with renal tumor(s)
* Subject will undergo a robot assisted partial nephrectomy
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for kidney cancer by this surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Post-operative complications evaluated according to the Clavien criteria | From surgery until 1 year of follow up
  Per and post-operative transfusion rates
Post-operative complications evaluated according to the Clavien criteria | From surgery until 1 year of follow up
  Medical or surgical complication rates
Post-operative complications evaluated according to the Clavien criteria | From surgery until 1 year of follow up
  Clavien's grading
Post-operative complications evaluated according to the Clavien criteria | From surgery until 1 year of follow up
  Urinary fistula rate
Post-operative complications evaluated according to the Clavien criteria | From surgery until 1 year of follow up
  Necessity for nephrectomy or re-exploration
Post-operative complications evaluated according to the Clavien criteria | From surgery until 1 year of follow up
  Length of hospital stay

SECONDARY OUTCOMES:
Renal function after robotic partial nephrectomy measured by biological parameters | Follow-up during 12 months
  Creatininemia
Renal function after robotic partial nephrectomy measured by biological parameters | Follow-up during 12 months
  MDRD GFR
Per-operative modalities of haemostasis procedure | At Surgery
  Haemostasis procedure
Per-operative modalities of haemostatic agent | At Surgery
  Haemostatic agent

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe BERNHARD, PHU, Principal Investigator — University Hospital, Bordeaux
Locations (15):
- France (15):
  - CHU Bordeaux, Bordeaux
  - CHU Grenoble, La Tronche
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - HCL Lyon, Lyon
  - CH Diaconesses, Paris
  - CHU La Pitié Salpétrière/ Kremlin Bicêtre, Paris
  - CH Saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Henri MONDOR, Paris
  - CHU Rennes - Centre Eugène Marquis, Rennes
  - CHU Strasbourg, Strasbourg
  - CH Foch, Suresnes
  - CHU Toulouse - Centre Claudius Régaud, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Margue G, Ingels A, Bensalah K, Doumerc N, Vaessen C, Roupret M, Audenet F, Mejean A, Bruyere F, Olivier J, Baumert H, Michel C, Paparel P, Parier B, Sebe P, Long JA, Lang H, Lebret T, Patard JJ, Bernhard JC. Late complications and 5 years outcomes of robotic partial nephrectomy in France: prospective assessment in the French Kidney Cancer Research Network (UroCCR 10). World J Urol. 2023 Aug;41(8):2281-2288. doi: 10.1007/s00345-023-04491-z. Epub 2023 Jul 6. PMID 37407720